CLINICAL TRIAL: NCT05460364
Title: A Randomized, Open-label, Multiple-dose, 6-sequence, 3-treatment, 3-period, Crossover Study to Evaluate the Pharmacokinetic Interaction and Safety Between BR1018-1 and BR1018-2 in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Pharmacokinetic Interaction and Safety Between BR1018-1 and BR1018-2 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: BR-FAEAC-CT-101
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Hypertension; Hyperlipidemia (E.G., Hypercholesterolemia)
MeSH Terms: conditions — Hypertension; Hyperlipidemias; Hypercholesterolemia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Sequence 1 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 1: A-B-C
  Interventions: Drug: BR1018-1; Drug: BR1018-2
- Sequence 2 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 2: A-C-B
  Interventions: Drug: BR1018-1; Drug: BR1018-2
- Sequence 3 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 3: B-A-C
  Interventions: Drug: BR1018-1; Drug: BR1018-2
- Sequence 4 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 4: B-C-A
  Interventions: Drug: BR1018-1; Drug: BR1018-2
- Sequence 5 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 5: C-A-B
  Interventions: Drug: BR1018-1; Drug: BR1018-2
- Sequence 6 (Experimental): The Investigational products will be administered according to the treatment groups(A,B,C) assigned to each sequence group in Period 1, Period 2, and Period 3.
  *sequence 6: C-B-A
  Interventions: Drug: BR1018-1; Drug: BR1018-2

INTERVENTIONS:
Drug: BR1018-1 — Treatment group A : One tablet of BR1018-1 administered alone once daily for 9 days.
  Treatment group C : One tablet each of BR1018-1 and BR1018-2 administered in combination once daily for 9 days.
Drug: BR1018-2 — Treatment group B : One tablet of BR1018-2 administered alone once daily for 9 days.
  Treatment group C : One tablet each of BR1018-1 and BR1018-2 administered in combination once daily for 9 days.

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic characteristics and compare the safety and tolerability after repeated separate or combined administrations of BR1018-1 and BR1018-2 in healthy adults.

DETAILED DESCRIPTION:
A total of 36 subjects will be randomized into 6 sequence groups, 6 subjects per sequence group. The Investigational Products wil be according to the treatment group (A,B,C) assigned to each sequence group in Period 1, Period 2 and Period 3.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged 19 to 55 years at screening
2. Those who weigh at least 50 kg at the time of screening and have a calculated body mass index (BMI) within the range of 18.0 to 30.0 kg/m2
3. Those who have been determined to be eligible as subjects through physical examinations and interviews conducted in accordance with this protocol. In other words, those who have no congenital or chronic diseases and have no abnormal symptoms or findings based on medical examination results within the last 3 years
4. Those who have been determined to be eligible as subjects as a result of clinical laboratory tests and electrocardiography performed according to this protocol (if the results are within the reference values of Inha University Hospital or if the investigator determines that the clinical laboratory test and electrocardiography results are not clinically significant even if they are out of range)
5. Those who voluntarily decide to participate in the study and provide written consent to follow the study directions after listening to and fully understanding the detailed explanation on this study

Exclusion Criteria:

1. Those who have clinically significant diseases associated with the cardiovascular system, respiratory system, liver, kidney, nervous system, endocrine system, blood/tumor, psychiatric disorders, or urinary system, as well as drug abuse, or a history thereof.
2. Those who have hypersensitivity reactions to drugs containing fimasartan, amlodipine, ezetimibe, atorvastatin, or same-class ingredients, yellow no. 5 (sunset yellow FCF), dihydropyridine derivatives, or to other drugs (aspirin, antibiotics, etc.), or a history of clinically significant hypersensitivity reactions thereto.
3. Those who have a hereditary disorder including galactose intolerance, Lapp lactase deficiency, glucose-galactose malabsorption, etc.
4. Those who have a history of gastrointestinal diseases (e.g., Crohn's disease, ulcerative disease, etc.) or gastrointestinal surgery (however, simple appendectomy or hernia repair are excluded) that may affect the absorption of drugs
5. Those who have clinically significant hypotension (systolic blood pressure ≤ 90 mmHg) or hypertension (systolic blood pressure ≥ 150 mmHg or diastolic blood pressure ≥ 95 mmHg) at screening
6. Those who show any of the following results in the screening tests

   * AST or ALT > 2 times the upper limit of the normal range
   * Total bilirubin > 2.0 mg/dL
   * CK > 2 times the upper limit of the normal range
   * Estimated glomerular filtration rate (eGFR) < 60 mL/min/1.73 m2
7. Those who continue to drink alcohol (>21 units/week; 1 unit = 10 g = 12.5 mL of pure alcohol), or who are unable to abstain from drinking during the clinical study period
8. Those who continue to smoke (>10 cigarettes/day), or who are unable stop smoking during hospitalization within the clinical study period
9. Those who have participated in another clinical study or bioequivalence test (the last day of administration of the investigational product or bioequivalence test drug) within 6 months prior to the first administration date
10. Those who have donated whole blood within 60 days prior to the first day of administration or donated blood components within 30 days prior to the first day of administration or who have received a blood transfusion within 30 days
11. Those who took any prescription drugs or herbal medicines within 14 days prior to the first day of administration or any over-the-counter (OTC) drugs within 7 days prior to the first day of administration (however, if other conditions are appropriate according to the judgment of the investigator, they may participate in the clinical study.)
12. Those who took drugs inducing and inhibiting drug-metabolizing enzymes, such as barbiturates, within 30 days prior to the study initiation
13. Those who have been on a diet (especially grapefruit juice or its products) that may affect the absorption, distribution, metabolism, and excretion of the drug within 7 days prior to the first day of administration
14. Pregnant women, potentially pregnant women, or breast-feeding women
15. Those who do not agree to rule out the possibility of their and their spouses' or sexual partners' pregnancy by using medically acceptable methods of contraception* throughout the entire period from the date of the first administration of the investigational product to the end of the clinical study

    * Medically acceptable methods of contraception: Combined use of intrauterine device, vasectomy, tubal ligation, and barrier methods (male condom, female condom, cervical cap, diaphragm, sponge, etc.) or combined use of two or more barrier methods if spermicide is used
16. Those who are unwilling or unable to comply with the dietary and lifestyle guidelines required for the clinical study
17. Those who have clinically significant abnormalities in the results of other clinical laboratory tests or who have been determined by the investigator to be ineligible to participate in the clinical study due to other reasons (e.g., non-compliance with instructions, uncooperative attitude, etc.)

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-08-04 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

PRIMARY OUTCOMES:
AUC0-24,ss | 0-48 hours after administration
  Area under the plasma drug concentration-time curve from 0 to time t of BR1018-1 and BR1018-2
Cmax,ss | 0-48 hours after administration
  Maximum concentration of drug in plasma of BR1018-1 and BR1018-2

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No